CLINICAL TRIAL: NCT02386111
Title: A Phase l/ll Study of Varlilumab in Combination With Sunitinib in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: A Study of Varlilumab (Anti-CD27) and Sunitinib in Patients With Metastatic Clear Cell Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio re-prioritization
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDX1127-04
Record Dates: First submitted 2015-03-06; First posted 2015-03-11 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell; Kidney Diseases; Kidney Neoplasms; Urogenital Neoplasms; Urologic Diseases; Urologic Neoplasms; Neoplasms; Neoplasms by Histologic Type; Clear-cell Metastatic Renal Cell Carcinoma
Keywords: Sutent
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Diseases; Kidney Neoplasms; Urogenital Neoplasms; Urologic Diseases; Urologic Neoplasms; Neoplasms; Neoplasms by Histologic Type; Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varlilumab and Sunitinib (Experimental)
  Interventions: Drug: Combination of varlilumab and sunitinib

INTERVENTIONS:
Drug: Combination of varlilumab and sunitinib — During the treatment phase of the study, eligible patients will receive varlilumab for up to 8 cycles. Treatment cycles are 6 weeks each with varlilumab administered once every 3 weeks and sunitinib administered daily for 4 weeks followed by a 2 week rest. There is no limit on the number of cycles of sunitinib. Patients may be discontinued from receiving study treatment (sunitinib or varlilumab) based on the results of disease assessments or if experiencing side effects that make study therapy intolerable.
  Phase l Dose: The planned dose of varlilumab will be dependent on the cohort assigned at enrollment. Varlilumab doses are 0.3 mg/kg, 1 mg/kg or 3 mg/kg.
  The Study was terminated prior to initiation of Phase II.
  All patients will receive sunitinib at a dose of 50 mg.

SUMMARY:
This is a study to determine the clinical benefit (how well the drug works), safety, and tolerability of combining varlilumab and sunitinib. The study will enroll patients with metastatic clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
Varlilumab is a fully human monoclonal antibody that binds to a molecule called CD27 found on certain immune cells and may act to promote anti-tumor effects.

Sunitinib is a small molecule that inhibits multiple receptor tyrosine kinases (RTKs) some of which play a role in tumor growth and progression of cancer.

This study will evaluate the safety, tolerability and efficacy of the anti-CD27 antibody varlilumab in combination with sunitinib.

Eligible patients that enroll in the dose escalation portion of the study will be assigned to one of three dose levels of varlilumab in combination with 50 mg of sunitinib. The first phase of the study will test the safety profile of the combination and determine which dose of varlilumab will be studied in Phase ll* of the overall study.

*Note: This Study was terminated prior to initiation of Phase II.

All patients enrolled in the study will be closely monitored to determine if there is a response to the treatment as well as for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of predominant clear cell renal cell carcinoma.
2. Advanced metastatic disease
3. Documented progressive disease based on radiographic, clinical or pathologic assessment during or subsequent to last therapy.
4. For Phase l, no more than 3 prior anticancer regimens (IL-2 or interferon do not count towards the total).
5. Measurable (target) disease.
6. Life expectancy ≥ 12 weeks.
7. If of childbearing potential (male or female), agrees to practice an effective form of contraception during study treatment and for at least 70 days following last treatment dose.
8. Must have available tumor tissue and consent to biopsy while on study.

Exclusion Criteria:

1. Prior therapy with an anti-CD27 antibody.
2. Previous treatment with sunitinib.
3. Use of any experimental immunotherapy.
4. Chemotherapy within 21 days or at least 5 half-lives (whichever is shorter) prior to the planned start of study treatment.
5. Systemic radiation therapy within 4 weeks, prior focal radiotherapy within 2 weeks, or radiopharmaceuticals (strontium, samarium) within 8 weeks prior to the first dose of study treatment.
6. Use of immunosuppressive medications within 4 weeks or systemic corticosteroids within 2 weeks prior to first dose of study treatment.
7. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
8. Active, untreated central nervous system metastases.
9. Active autoimmune disease or a documented history of autoimmune disease.
10. Active diverticulitis.
11. Significant cardiovascular disease including CHF or poorly controlled hypertension.
12. Impairment of gastrointestinal function or gastrointestinal disease that may alter the absorption of sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Phase 1: Safety and tolerability of varlilumab and varlilumab in combination with sunitinib as measured by incidence of drug related adverse events (AEs), serious drug related AEs, dose-limiting toxicities and laboratory test abnormalities. | Safety follow-up is 100 days from last study drug dose.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Helen Diller Comprehensive Cancer Center, San Francisco, California
  - George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania